CLINICAL TRIAL: NCT03644563
Title: Impacting the Oral HPV Continuum: MOUTH Study (Men and Women Offering Understanding of Throat HPV)
Brief Title: Men and Women Offering Understanding of Throat HPV
Acronym: MOUTH
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00119537; R35DE026631 (NIH)
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Oropharyngeal Cancer; Human Papilloma Virus
Keywords: Oral HPV; Persistent infection; Oropharyngeal cancer (OPC); HPV antibody; HPV Screening Study
MeSH Terms: conditions — Oropharyngeal Neoplasms; Persistent Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Oral rinse sample: a sample of oral exfoliated cells will be collected using 10 mL of saline.Oral rinse samples will be tested for HPV DNA and/or RNA.
  Saliva sample: Saliva sampling kits designed to preserve HPV (OraGene RNA kit from DNA Genotek) will be used to collect oral samples from all participants.
  Urine sample: Urine will be tested for HPV DNA as a surrogate for genital HPV infection.
  Blood collection: Each sample will be tested for HPV antibodies. Capsid antibodies will be measured using virus like particle-based ELISA assays. Antibodies to the E6 and E7 proteins will be measured in a glutathione capture ELISA assays.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Follow-up: Those subjects with oncogenic oral HPV infection and/or HPV oncogene serum antibodies from screening.

SUMMARY:
This study will screen people for oncogenic oral Human Papillomavirus (HPV) infection and antibodies to form a cohort of people who may be at increased risk of HPV-oropharyngeal cancer (HPV-OPC). The investigators will follow these individuals prospectively to evaluate oncogenic oral HPV persistence, risk factors, and biomarkers for persistence.

DETAILED DESCRIPTION:
This study will provide one of the first estimates of long-term oral HPV natural history, and the effect of biologic and behavioral risk factors, including HIV, on this natural history. Phase 1 of the study will screen approximately 1500 people for oncogenic oral HPV biomarkers. Phase 2 of the study will follow only those subjects with oncogenic oral HPV infection and/or HPV serum oncogene antibodies from Phase 1 (and those previously identified as having oncogenic oral HPV infection in a previous study) with annual follow-up for oncogenic oral HPV persistence.

Understanding persistent oncogenic oral HPV infection is the focus of this study. Understanding which factors drive oral HPV infection to become persistent or progress to malignancy is critical to determine who is at high risk for oropharyngeal cancer and may benefit from screening and prevention. It is presumed that persistent oncogenic oral HPV infections are necessary for progression to HPV-OPC.

The study is led by Dr. Amber D'Souza and Dr Carole Fakhry (Johns Hopkins) and participants are being enrolled in Baltimore MD (Johns Hopkins) and in New York (Mt. Sinai).

ELIGIBILITY:
Participants in the Phase 1 Screening

Inclusion criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* 18 and older (enrollment at most sites will be restricted to 30 and older since this demographic has the highest prevalence of infection; however, individuals and/or partners of someone with an HPV-related cancer, for example, are at increased risk so will be enrolled in the larger age range).
* Willing to be contacted to arrange follow-up visits, if determined to be eligible for phase 2
* Ability to understand and the willingness to sign a written informed consent document

In addition, individuals must meet at least one of the following criteria:

* Male, aged 30 and older, with 2 or more lifetime oral sex
* History of anal or genital dysplasia or cancer
* Partners of someone with an HPV-related cancer (HPV-positive OPC, anal cancer or genital cancer)
* Known oncogenic HPV-positive biomarker from prior studies or testing, regardless of number of partners.

Exclusion criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Presence of medical or psychiatric condition affecting ability to give voluntary, informed consent.
* Participants who do not speak English cannot enroll because the consent and study survey are only available in English. However, if there is a hearing, literacy or minor fluency issue and the participant requests assistance from a family member or the study coordinator, this individual may still enroll and receive this assistance to ensure they fully hear and understand everything being asked.
* History of head and neck cancer

Participants in the Phase 2 Follow-Up

Inclusion criteria:

* Oncogenic oral HPV infection and/or HPV serum oncogenic antibodies detected in phase 1
* Willingness to complete annual follow up visits

Exclusion criteria:

• Unable to complete annual follow up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Target sample size: 1325 (phase 1), ~250 (phase 2) Inclusion of women and minorities: Primary enrollment is restricted to men, given their higher risk of infection (see eligibility criteria). However, the investigators expect to enroll women with cervical dysplasia and partners of patients with HPV-related cancer (~125 expected women enrollees). Enrollment is across many different sources (geographically, and by clinic type), and is inclusive of diverse racial and ethnic backgrounds. Enrollment is not stratified by race but the investigators expect to enroll at least 175 minorities in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Oncogenic oral HPV infection present or absent in oral rinse sample | Baseline to end of four year follow-up and data abstraction/linkage.
  To explore the effects of biologic (microbiome, oral immune response, biologic sex) risk factors for oncogenic oral HPV persistence

SECONDARY OUTCOMES:
HPV16 E6 antibodies present or absent in serum sample | Baseline to end of four year follow-up and data abstraction/linkage.
  To explore whether E6 and E7 seropositivity (to HPV16 or any oncogenic HPV) are markers for oncogenic oral HPV persistence among high-risk groups

CONTACTS AND LOCATIONS:
Overall Officials: Amber D'Souza, PhD, Principal Investigator — Bloomberg Johns Hopkins School of Public Health
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] D'Souza G, Clemens G, Troy T, Castillo RG, Struijk L, Waterboer T, Bender N, Pierorazio PM, Best SR, Strickler H, Wiley DJ, Haddad RI, Posner M, Fakhry C. Evaluating the Utility and Prevalence of HPV Biomarkers in Oral Rinses and Serology for HPV-related Oropharyngeal Cancer. Cancer Prev Res (Phila). 2019 Oct;12(10):689-700. doi: 10.1158/1940-6207.CAPR-19-0185. Epub 2019 Aug 16. PMID 31420362
- [Result] D'Souza G, Tewari SR, Troy T, Waterboer T, Struijk L, Castillo R, Wright H, Shen M, Miles B, Johansson M, Robbins HA, Fakhry C. Prevalence of oral and blood oncogenic human papillomavirus biomarkers among an enriched screening population: Baseline results of the MOUTH study. Cancer. 2023 Aug 1;129(15):2373-2384. doi: 10.1002/cncr.34783. Epub 2023 Apr 9. PMID 37032449
- [Result] D'Souza G, Tewari SR, Troy T, Webster-Cyriaque J, Wiley DJ, Lahiri CD, Palella FJ, Gillison ML, Strickler HD, Struijk L, Waterboer T, Ho K, Kwait J, Lazar J, Weber KM, Fakhry C. Oncogenic Oral Human Papillomavirus Clearance Patterns over 10 Years. Cancer Epidemiol Biomarkers Prev. 2024 Apr 3;33(4):516-524. doi: 10.1158/1055-9965.EPI-23-1272. PMID 38294704
- See also: MOUTH Study Website — http://bit.ly/MOUTHStudy